CLINICAL TRIAL: NCT02676557
Title: The Lamina Cribrosa (LC) Morphologic Changes in the Eyes After Laser-Assisted in Situ Keratomileusis (LASIK)
Brief Title: The Lamina Cribrosa (LC) Changes in the Eyes After Laser-Assisted in Situ Keratomileusis (LASIK)
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Changwon Kee, Professor, Samsung Medical Center
Other Study IDs: LASIK-LC study
Record Dates: First submitted 2015-10-19; First posted 2016-02-08 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: The Lamina Cribrosa and Optic Nerve Head Changes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- LASIK
  Interventions: Device: Exposed to the high pressure during the surgery

INTERVENTIONS:
Device: Exposed to the high pressure during the surgery

SUMMARY:
The burden of LASIK surgery on optic nerve head (ONH) has been controversial. Until now, the change of retinal nerve fiber layer (RNFL) thickness was used as the indicator of the study. In the present study, the investigators intended to investigate whether the changes of the deep and superficial structures around ONH exist or not using EDI OCT.

ELIGIBILITY:
Inclusion Criteria:

* the myopic patients who were supposed to undergo LASIK surgery in the Samsung Medical Center

Exclusion Criteria:

* Optic nerve head abnormalities at preoperative examination
* Previous ocular surgical history

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The myopic patients who were supposed to undergo LASIK surgery
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-04; Primary Completion 2014-08 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change of lamina cribrosa (LC) depth | before the surgery, postoperative 1 day, 1 week, 1 month, and 3 months
  micro millimeter
Change of lamina cribrosa (LC) thickness | before the surgery, postoperative 1 day, 1 week, 1 month, and 3 months
  micro millimeter
Change of optic nerve head (ONH) width | before the surgery, postoperative 1 day, 1 week, 1 month, and 3 months
  micro millimeter

SECONDARY OUTCOMES:
Change of optic nerve head minimum rim width | before the surgery, postoperative 1 day, 1 week, 1 month, and 3 months
  micro millimeter